CLINICAL TRIAL: NCT01166022
Title: Randomized, Controlled Clinical Trial of Exercise in Patients With Spinal Muscular Atrophy (SMA)
Brief Title: Clinical Trial of Exercise in Patients With Spinal Muscular Atrophy (SMA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Darryl C. De Vivo, Sidney Carter Professor of Neurology and Professor of Pediatrics, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAE8200; A-15886 (Other: CU)
Record Dates: First submitted 2010-07-14; First posted 2010-07-20 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Spinal Muscular Atrophy; Neuromuscular Disease
Keywords: Spinal Muscular Atrophy; Exercise; Conditioning; Strengthening
MeSH Terms: conditions — Muscular Atrophy, Spinal; Neuromuscular Diseases; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Experimental): Muscle strengthening program using weights and resistance bands in combination with a home based cycle ergometry program. The home-based exercise program will be performed up to 5 times weekly.
  Interventions: Other: Exercise
- Typical Activity (No Intervention): Subjects in this group will be asked to maintain their typical daily activity. Those assigned to this arm will be given the opportunity to join the intervention arm seven months after their screening visit.

INTERVENTIONS:
Other: Exercise — Muscle strengthening program using hand weights and resistance bands in combination with a home based cycle ergometry. This home-based exercise program will be performed up to 5 times weekly. Each session will consist of up to 30 minutes of cycling and 30 minutes of strengthening.
  Arms: Exercise

SUMMARY:
This study is being conducted to test whether exercise can be effectively used as an intervention to treat Spinal Muscular Atrophy (SMA). In order to answer this question, the investigators will enroll 14 subjects with SMA between ages 8 and 50 and ask them to complete an 18 month training schedule. At some points subjects will be asked to closely follow a specific training regimen and at other points they may be asked to exercise in the same manner they do normally. The exercises they will be asked to perform include biking on a stationary cycle and lifting hand weights. Subjects will be asked to come in to the clinic seven times over the course of the study to perform tests. These tests include motor function measures, a physical exam, questionnaires, a exercise capacity test which involves riding a stationary bicycle, and test where the subject is asked to walk as far as they can in six minutes. The main goal of the study is to see if the subjects who participate in the exercise protocol have larger increases in the distance they can walk in six minutes than those who do not.

ELIGIBILITY:
Inclusion Criteria:

1. Weakness and hypotonia consistent with the clinical diagnosis of SMA type 3, i.e. having achieved the ability to walk independently
2. Laboratory documentation of homozygous absence of SMN1 exon 7
3. ability to walk at least 25 meters without assistance
4. Aged 8 to 50 years at the time of enrollment
5. Ability to tread the stationary cycle ergometer
6. Written informed consent of patient (if ≥ 18 years of age) or parents/guardian (if < 18 years of age), and assent for participants who are of minor age.

Exclusion Criteria:

1. Inability to walk independently at least 25 meters
2. Any acute co-morbid condition interfering with study participation in the judgment of the investigators within 7 days of enrollment including bacterial infection, viral infectious process, food poisoning, temperature > 99.0ºF, need for acute treatment or observation due to any other reason, as judged by the investigator; patient can be included after resolution of the acute event
3. Use of investigational medications intended for the treatment of SMA including riluzole, valproic acid, hydroxyurea, oral use of albuterol, sodium phenylbutyrate, butyrate derivatives, creatine, carnitine, growth hormone, anabolic steroids, or agents with known or presumed histone deacetylase (HDAC) inhibition, within 30 days prior to study entry. After signing informed consent, participants may discontinue prohibited medications and will then qualify for a screening visit after the 30 day wash-out period
4. Inability to meet study visit requirements, or cooperate reliably with functional testing and exercise protocol
5. Coexisting medical conditions that contraindicate travel, testing or moderate intensity exercise
6. Pregnant or breastfeeding women, or those intending to become pregnant during the course of the study.

Ages: 8 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2010-12; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Distance walked in the Six Minute Walk Test (6MWT). | Up to 19 months

CONTACTS AND LOCATIONS:
Overall Officials: Darryl C De Vivo, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University SMA Clinical Research Center, New York, New York, United States

REFERENCES:
- See also: Related Info — http://www.columbiasma.org